CLINICAL TRIAL: NCT03591952
Title: Gravity- Versus Suction-driven Large Volume Thoracentesis: a Randomized Controlled Study
Brief Title: Gravity- Versus Suction-driven Large Volume Thoracentesis
Acronym: GRAVITAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Fabien Maldonado, Associate Professor of Allergy/Pulmonary & Critical Care Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 180339; 180339 (Other: Vanderbilt University Medical Center)
Record Dates: First submitted 2018-06-11; First posted 2018-07-19 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Pleural Effusion
Keywords: Thoracentesis
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be randomly allocated into intervention (gravity-driven) and control (suction-driven) groups by opening an opaque study envelope just prior to starting the procedure containing group assignment. Participants will be blinded to the use of gravity VS. suction drainage to prevent knowledge of their group assignment from biasing their pain assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suction (Active Comparator): The pleural fluid will be drained by the syringe system with a one-way valve tubing system provided in the kit. Selection of the vacuum pressure will be at the discretion of the proceduralist, as per standard of care.
  Interventions: Procedure: Suction-Driven Thoracentesis
- Gravity (Experimental): The pleural fluid will be drained using gravity drainage to a bag positioned approximately 100 cm (approximately 40 inches) below the catheter entry point (see picture below) using the 40 inch tubing provided in the thoracentesis kit (CareFusion or Arrow).
  Interventions: Procedure: Gravity-Driven Thoracentesis

INTERVENTIONS:
Procedure: Suction-Driven Thoracentesis — Thoracentesis is a procedure in which a needle is inserted into the pleural space between the lungs and the chest wall. This procedure is done to remove excess fluid, known as a pleural effusion, from the pleural space to help one breathe easier.
  Arms: Suction
Procedure: Gravity-Driven Thoracentesis — Thoracentesis is a procedure in which a needle is inserted into the pleural space between the lungs and the chest wall. This procedure is done to remove excess fluid, known as a pleural effusion, from the pleural space to help one breathe easier.
  Arms: Gravity

SUMMARY:
Thoracentesis is a very common procedure, rarely associated with severe complications. One relatively common complication is chest discomfort, which is most of the time felt to be secondary to negative pleural pressures generated during the procedure. While most proceduralists use suction to drain the pleural fluid, some drain effusions by gravity only. The investigators propose to evaluate whether gravity-driven thoracentesis results in less discomfort for patients than suction-drive thoracentesis.

DETAILED DESCRIPTION:
Therapeutic thoracentesis aims to drain fluid from the pleural space to alleviate breathlessness. The amount of and speed with which the fluid can be safely drained in one setting is unclear, and likely depends on the physiology of the pleural effusion. The principle concern when draining a large amount of fluid quickly from the pleural space is that excessively negative pleural pressure may be generated; this occurs if the lung is unable to freely re-expand into the space previously occupied by fluid. Excessively negative pleural pressure and the resulting high transpulmonary pressure gradient are thought to be associated with several complications, including pneumothorax ex vacuo, chest discomfort, and re-expansion pulmonary edema (REPE). Evidence suggests that monitoring pleural pressures during thoracentesis via manometry does not mitigate this problem. In fact, data shows that whether manometry is used or not, most patients do experience clinically significant increase in chest discomfort during thoracentesis. Current methods for draining the pleural fluid include suction- (via vacuum bottles, wall suction or the use of large syringes with a one-way valve tubing system) or gravity-driven thoracentesis. Pressures generated by all suction techniques range from -200 to -500 cmH2O, and far exceed what are considered safe pleural pressures. Accordingly, in case of non-expandable lung, excessively negative pressures may develop quickly, exposing patients to complications. Some clinicians advocate for gravity drainage, which generates less negative pressures in the pleural space (specifically defined as the vertical distance between the catheter and the drainage bag, generally around -50 to -100 cmH20). While this technique is considered standard of care by some as it is potentially more comfortable for patients, it is also likely associated with longer procedures, and is not generally favored by clinicians who in general prefer suction drainage, despite the possible higher risk of complications.The investigators propose to study the impact of gravity- versus suction-driven large volume therapeutic thoracentesis on the development of chest discomfort during the procedure, and consider as secondary endpoints: the duration of the procedure, the amount of pleural fluid drained, the rate of REPE, the rate of pneumothorax ex vacuo.

ELIGIBILITY:
Inclusion Criteria:

1. Referral to pulmonary services for large-volume thoracentesis
2. Presence of a symptomatic moderate or large free-flowing (non-septated) pleural effusion on the basis of:

   1. Chest radiograph: effusion filling ≥ 1/3 the hemithorax, OR
   2. CT-scan: maximum AP depth of the effusion ≥ 1/3 of the AP dimension on the axial image superior to the hemidiaphragm, including atelectatic lung completely surrounded by effusion, OR Ultrasound: effusion spanning at least three interspaces, with depth of 3 cm or greater in at least one interspace, while the patient sits upright.
3. Age > 18

Exclusion Criteria:

1. Inability to provide informed consent
2. Patient has already been enrolled in this study
3. Study subject has any disease or condition that interferes with safe completion of the study including:

   1. Coagulopathy, with criteria left at the discretion of the operator
   2. Hemodynamic instability with systolic blood pressure <90 mmHg or heart rate > 120 beats/min, unless deemed to be stable with these values by the attending physicians
4. Pleural effusion is smaller than expected on bedside pre-procedure ultrasound
5. Referral is for diagnostic thoracentesis only
6. Presence of more than minimal septations and/or loculations on bedside pre-procedure ultrasound
7. Inability to sit for the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Difference in post-procedure chest discomfort scores between control (suction) and intervention (gravity) groups | One-time assessment, 5 minutes after thoracentesis catheter is removed (on day 1)
  As measured in millimeters along a 10 cm Visual Analog Scale (VAS). The estimated minimal clinically important difference is 15 mm. Descriptive statistics including means, standard deviations, and ranges will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention versus (vs) control, will be made using the t-test or Wilcoxon Rank Sum test. Mixed model will be employed to assess the trend of pain score measured across pre-, intra-, and post-procedure.

SECONDARY OUTCOMES:
Incidence of pneumothorax | 20 minutes after thoracentesis catheter is removed (on day 1)
  Assessed as either present or absent on the immediate post-procedure chest radiograph per radiologist interpretation. Descriptive statistics including percentages and frequencies will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the Chi-square test.
Incidence of clinically-significant re-expansion pulmonary edema | 20 minutes after thoracentesis catheter is removed (on day 1)
  Assessed as present if immediate post-procedure chest radiograph demonstrates new pulmonary edema per radiologist interpretation when compared to pre-procedure radiograph in the hemithorax that underwent thoracentesis, and subject has post-procedure new-onset or worsened hypoxic respiratory failure. Descriptive statistics including percentages and frequencies will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the Chi-square test.
Incidence of radiographically-apparent re-expansion pulmonary edema | 20 minutes after thoracentesis catheter is removed (on day 1)
  Assessed as present if immediate post-procedure chest radiograph demonstrates new pulmonary edema per radiologist interpretation when compared to pre-procedure radiograph in the hemithorax that underwent thoracentesis. Descriptive statistics including percentages and frequencies will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the Chi-square test.
Volume of pleural fluid removed by the thoracentesis procedure | Immediately after the thoracentesis catheter is removed, on day 1
  Measured in milliliters. Descriptive statistics including means, standard deviations, and ranges will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the t-test or Wilcoxon Rank Sum test.
Improvement in dyspnea scores | From 1 minute pre-procedure to 5 minutes after thoracentesis catheter is removed (on day 1)
  Assessed in millimeters along a 10 cm Visual Analog Scale (VAS), from pre-procedure (baseline) to 5 minutes after completion of the procedure. Descriptive statistics including means, standard deviations, and ranges will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using either the t-test or Wilcoxon Rank Sum test.
Duration of procedure | During the procedure, on day 1, intraoperative
  Measured in seconds, assessed from the time the thoracentesis catheter is introduced to the time the catheter is removed. Descriptive statistics including means, standard deviations, and ranges will be presented. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity will be made. If necessary, data will be transformed using Box-Cox power transformation. Comparisons between groups, i.e. intervention vs control, will be made using the t-test or Wilcoxon Rank Sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Maldonado, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Lentz RJ, Shojaee S, Grosu HB, Rickman OB, Roller L, Pannu JK, DePew ZS, Debiane LG, Cicenia JC, Akulian J, Walston C, Sanchez TM, Davidson KR, Jagan N, Ahmad S, Gilbert C, Huggins JT, Chen H, Light RW, Yarmus L, Feller-Kopman D, Lee H, Rahman NM, Maldonado F; Interventional Pulmonary Outcomes Group. The Impact of Gravity vs Suction-driven Therapeutic Thoracentesis on Pressure-related Complications: The GRAVITAS Multicenter Randomized Controlled Trial. Chest. 2020 Mar;157(3):702-711. doi: 10.1016/j.chest.2019.10.025. Epub 2019 Nov 9. PMID 31711990